CLINICAL TRIAL: NCT06409351
Title: Multi-mOdal Training Program to Promote Physical actIVity After sTrokE: MOTIVATE
Brief Title: Multi-modal Training Program to Promote Physical Activity After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Singapore Institute of Technology (Other); National Neuroscience Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/2015; 06/FY2023/P1/21-A36 (Other Grant/Funding Number: National Neuroscience Institute of Singapore Pte Ltd (NNI))
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Stroke; Physical Inactivity
Keywords: Physical activity; Behavioural change; Implementation Science; Stroke
MeSH Terms: conditions — Stroke; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either treatment or control group only during the duration of the study
Who Masked: Outcomes Assessor
Masking Description: Only the outcomes assessor is masked. No other parties are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Study period: 6 months (1st 3 months intervention, last 3 months no intervention) No. of sessions: up to 6 per participant Mode: 3 sessions are conducted face-to-face and 3 sessions via telehealth methods e.g. phone, text message or video conferencing using virtual platforms like zoom.
  Where: Face-to-face at the participant's preferred exercise space like home, outdoor fitness zone, parks, gyms etc.
  Duration of sessions: each face-to-face session will take 60-90 mins Details of intervention: Physical activity counselling on adaptation of exercises, goal setting, action planning, problem solving around barriers to physical activity and provision of study resources
  Interventions: Behavioral: Intervention group
- Control group (Active Comparator): Study period: 6 months No. of sessions: 2 sessions (at month 1 and 3) Mode: Face-to-face Where: At the participant's home Duration of session: 20- 30 minutes Details of control: physical activity information without any other support.
  Interventions: Behavioral: Intervention group

INTERVENTIONS:
Behavioral: Intervention group — Please refer to arm descriptions
  Other Names: MOTIVATE

SUMMARY:
The goal of this study is to learn if a behavioral change intervention can improve physical activity in stroke survivors living in the community.

The main question it aims to answer is, if a behaviour change intervention and personalised physical activity prescription, are effective in improving the time spent in moderate to vigorous physical activity amongst chronic stroke survivors.

Researchers will compare the intervention group to a control group, to see if physical activity counselling and a personalized physical activity prescription is more effective in improving moderate to vigorous physical activity, than usual care alone. The study period for each participant is 6 months. Assessments are conducted at month 1 (baseline), 3 and 6.

The control group will receive only usual care, which consists of an information sheet on physical activity with the following content: (1) Why be active and (2) How to be active (with URL links to resources and videos). The usual care is delivered at 3-time points during month 1, 3 and 6.

The intervention group will receive usual care and a behavioral change intervention. The behavioral change intervention consists of up to 6 individual physical activity counselling sessions and a personalized physical activity prescription. The 6 sessions will take place only during months 1 to 3 and there will be no intervention during months 4 to 6. Of the 6 sessions, 3 are conducted face-to-face and another 3 sessions will take place using telehealth methods such as phone, text messaging and videoconference. Participants can meet the study physiotherapist at their preferred exercise space during the 3 face-to-face sessions. The physical activity counselling sessions consist of goal setting and action planning, and problem-solving barriers around participation in physical activity. The overall aim is to increase time spent in moderate-vigorous physical activity.

DETAILED DESCRIPTION:
The MOTIVATE study will take place in Singapore with participants recruited through hospital-based stroke clinics, rehabilitation facilities, and stroke support organizations via posters, email, word of mouth, and social media. Potential participants can sign up by self-registering on the study URL link or through referrals from healthcare professionals and study members. Participants will be screened for eligibility via telephone using the inclusion and exclusion criteria and the Get Active Questionnaire. Participants. Those who have not engaged in regular exercise are required to obtain medical clearance. Informed consent will be taken by a study team member.

This trial will use a 1:1 concealed randomisation, to allocate participants with chronic stroke to an intervention group (n= 60) or control group (n = 60). Between-group comparisons will be made at 3 time points: months 1, 3 and 6.

The control group will receive usual care, which consists of 3 face-to-face sessions on general physical activity recommendations, lasting 30 to 60 minutes each during months 1, 3, and 6. Participants will be given an information sheet on the importance and benefits of physical activity after a stroke and general guidelines on how to start to be active. The general guidelines on how to be active include engaging in 150 minutes of moderate-intensity physical activity per week. The information sheet will also include links to publicly accessible online resources.

The intervention group will receive a behavioural change intervention, in addition to usual care. Information sheet about general guidelines on physical activity will be handed to the intervention group, as per control group. Each participant will receive up to 6 sessions of tailored behavioural change intervention during months 1 to 3 and there will be no intervention during months 4 to 6. Of the 6 sessions, 3 are face-to-face and another 3 will take place using telehealth methods such as phone, text messaging and videoconference. The tailoring of the intervention allows participants to decide the location during face-to-face sessions, how many sessions and how the sessions are spaced out during the 3-month intervention period and which sessions are face-to-face or telehealth. The preferred meeting location may include exercise spaces within home, common spaces just outside their homes and under their housing blocks, outdoor fitness zones or parks near home and residential or inclusive public gyms. The behavioural change intervention consists of physical activity counselling and prescription of a personalized physical activity plan. The first session will be conducted in-person, to allow the study physiotherapist to identify the participant's physical function, safety concerns and the impact of medical, social, environmental and resources on mobility. During the initial visit, the venue, frequency and mode of support (face-to-face or virtual) for subsequent sessions will be established. The study physiotherapist will provide physical activity counselling, set goals and discuss action plans to enhance moderate intensity physical activity, problem solve barriers on physical activity and prescribe a personalized physical activity plan. Subsequent sessions can include (1) training on physical activity modification to accommodate the weak arm and / leg at the participant's preferred exercise location, (2) taking videos of the personalized adapted exercises using the participant's phone when meeting face-to-face and (3) in-person or virtual support sessions to review physical activity progress and action plans.

A process and cost-utility evaluation will be embedded into the study design and conducted concurrently.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 years and over
* Haemorrhagic or ischaemic stroke
* At least 6 months post-stroke
* Living at home
* Able to walk independently +/- gait aid short distances (self-reported)
* Have sufficient cognition and/or carer support to engage in the interventions (clinical judgement)
* Agreement to undertake a supported self-management physical activity intervention programme

Exclusion Criteria:

* Living in residential care
* Unstable cardiac conditions, severe arthritis, or other conditions limiting the ability to exercise
* Advised by GP/consultant not to undertake moderate-intensity exercise for health reason
* Currently already participating in physical activity that meets recommended levels (150mins of moderate-vigorous physical activity)
* Enrolled in another physical activity intervention trial

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Duration of moderate to vigorous physical activity | Initial assessment (month 1), month 3 and 6 follow-up.
  Average minutes/day, measured by Fitbit Inspire 3 tracker

SECONDARY OUTCOMES:
Number of steps per day | Initial assessment (month 1), month 3 and 6 follow-up.
  Number of steps per day, measured by Fitbit Inspire 3 tracker
International Physical Activity Questionnaire Short Form (IPAQ-SF) | Initial assessment (month 1), month 3 and 6 follow-up.
  Duration (in minutes) and frequency (days) of walking, moderate-intensity, and vigorous-intensity activity, which are used to compute the total score.
Modified Rankin Scale | Initial assessment (month 1), month 3 and 6 follow-up.
  0. No symptoms
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability: unable to carry out all previous activities but able to look after own affairs without assistance
  3. Moderate disability: requiring some help, but able to walk without assistance
  4. Moderately severe disability: unable to walk without assistance, and unable to attend to own bodily needs without assistance
  5. Severe disability: bedridden, incontinent, and requiring constant nursing care and attention
  Outcome data: One score from a 6-point scale of 0-5.
Functional Ambulation Category | Initial assessment (month 1), month 3 and 6 follow-up.
  0) Patient cannot walk, or needs help from 2 or more persons
  1. Patients needs firm continuous support from 1 person who helps carrying weight and with balance
  2. Patient needs continuous or intermittent support of one person to help with balance and coordination
  3. Patient requires verbal supervision or stand-by help from one person without physical contact
  4. Patient can walk independently on level ground, but requires help on stairs, slopes or uneven surfaces
  5. Patient can walk independently anywhere
  Outcome data: One score from a 6-point scale of 0-5
Comfortable gait speed | Initial assessment (month 1), month 3 and 6 follow-up.
  Comfortable walking speed equals to predetermined distance divided by the average time taken from 2 trials to walk that distance comfortably or naturally (e.g., 5m/__sec).
Fast gait speed | Initial assessment (month 1), month 3 and 6 follow-up.
  Fast walking speed equals to predetermined distance divided by the average time taken from 2 trials to walk that distance as fast as possibly safe (e.g., 5m/__sec).
Life-space Assessment Measure | Initial assessment (month 1), month 3 and 6 follow-up.
  For the five "Life-Space Levels," each "Yes" is given a point value, starting with 1 (life-space level 1) and increasing by 1 point for each life-space level (2 for "Yes" in life-space level 2, 3 for "Yes" in life-space level 3, etc.).
  For frequency of each life-space level [less than 1 time per week (score = 1), 1-3 times per week (score = 2), 4-6 times per week (score = 3), or daily (score = 4)].
  For independence level, requiring assistance or use of any equipment [personal assistance (score = 1), equipment only (score = 1.5), or neither equipment nor personal assistance (score = 2)].
  Outcome data: The total score ranges from 0 ("totally bed-bound") to 120 ("traveling out of town every day without assistance").
Fall Efficacy Scale International (FES-I) | Initial assessment (month 1), month 3 and 6 follow-up.
  The Short FES-I consists of seven items
  Each item is scored on a 4-point scale:
  1. Not concerned at all
  2. Somewhat concerned
  3. Fairly concerned
  4. Very concerned
  Outcome data: Total score ranging from 7 (no concern about falling) to 28 (severe concern about falling).
Self-Efficacy for Exercise Scale (SEES) | Initial assessment (month 1), month 3 and 6 follow-up.
  Consists of 9 questions on the individual's confidence in their ability to engage in exercise. Each item is rated on a 11-point scale. Score of 0 indicates "not confident", and score of 10 indicates "very confident".
  Outcome data: Total score ranges from 0 ("not confident" in own ability to engage in exercise) to 90 ("very confident" in own ability to engage in exercise)
Fatigue Severity Scale - 7 item (FSS-7) | Initial assessment (month 1), month 3 and 6 follow-up.
  The FSS-7 consists of seven items, and the responses are scored on a seven-point scale, where 1 indicates "strongly disagree" and 7 indicates "strongly agree."
  Outcome data: Total score ranges from 7 to 49, with higher scores indicating more severe fatigue and greater impact on activities.
Fatigue screening tool (SF-CAT) | Initial assessment (month 1), month 3 and 6 follow-up.
  Yes/no screening questions to 16 questions that cover fatigue, mood, sleep quality, new / uncontrolled conditions, physical / nutrition status, role of medication consumption of alcohol, new / undiagnosed cognitive impairment, speech and language disorder.
Depression and Anxiety (PHQ-4) | Initial assessment (month 1), month 3 and 6 follow-up.
  The responses are scored on a four-point scale, where 0 indicates "not at all" and 3 indicates "nearly every day."
  Outcome data: Total score ranges from 0 to 12, with higher scores indicating greater severity of depression and anxiety symptoms.
Global Sleep Assessment Questionnaire (GSAQ) | Initial assessment (month 1), month 3 and 6 follow-up.
  Consists of 11 questions, rated on a 4-point scale ("never", "sometimes", "usually", "always").
  Outcome data: More "always" responses indicate better sleep quality.
EQ-5D | Initial assessment (month 1), month 3 and 6 follow-up.
  Outcome data: index values are used in the estimation of quality-adjusted life year (QALY) gains in economic analysis.
Global Rating of Change on Physical Activity and Fatigue | Month 3 and 6 follow-up.
  Score rated on a 15-point scale, ranging from -7 (a very great deal worse) to +7 (a very great deal better). A score of 0 indicates unchanged.
  Outcome data: One score from the 15-point scale.
Adapted Client Service Receipt Inventory (CSRI) | Initial assessment (month 1), month 3 and 6 follow-up.
  Cost estimate of resource utilization to generate an average cost per participant

CONTACTS AND LOCATIONS:
Overall Officials: Shamala Thilarajah, PhD, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
The study protocol with the statistical analysis plan will be published in a peer-reviewed journal.
Supporting Information: Study Protocol, SAP
Time Frame: To be published ahead of the completion of the trial
Access Criteria: The protocol will be available as per the publishing journal's options.

REFERENCES:
- [Background] Hardie K, Hankey GJ, Jamrozik K, Broadhurst RJ, Anderson C. Ten-year risk of first recurrent stroke and disability after first-ever stroke in the Perth Community Stroke Study. Stroke. 2004 Mar;35(3):731-5. doi: 10.1161/01.STR.0000116183.50167.D9. Epub 2004 Feb 5. PMID 14764929
- [Background] Turan TN, Nizam A, Lynn MJ, Egan BM, Le NA, Lopes-Virella MF, Hermayer KL, Harrell J, Derdeyn CP, Fiorella D, Janis LS, Lane B, Montgomery J, Chimowitz MI. Relationship between risk factor control and vascular events in the SAMMPRIS trial. Neurology. 2017 Jan 24;88(4):379-385. doi: 10.1212/WNL.0000000000003534. Epub 2016 Dec 21. PMID 28003500
- [Background] Fini NA, Bernhardt J, Said CM, Billinger SA. How to Address Physical Activity Participation After Stroke in Research and Clinical Practice. Stroke. 2021 Jun;52(6):e274-e277. doi: 10.1161/STROKEAHA.121.034557. Epub 2021 May 6. No abstract available. PMID 33951930
- [Background] WHO Guidelines on Physical Activity and Sedentary Behaviour. Geneva: World Health Organization; 2020. Available from http://www.ncbi.nlm.nih.gov/books/NBK566045/ PMID 33369898
- [Background] Billinger SA, Arena R, Bernhardt J, Eng JJ, Franklin BA, Johnson CM, MacKay-Lyons M, Macko RF, Mead GE, Roth EJ, Shaughnessy M, Tang A; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Lifestyle and Cardiometabolic Health; Council on Epidemiology and Prevention; Council on Clinical Cardiology. Physical activity and exercise recommendations for stroke survivors: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 Aug;45(8):2532-53. doi: 10.1161/STR.0000000000000022. Epub 2014 May 20. PMID 24846875
- [Background] Thilarajah S, Bower KJ, Pua YH, Tan D, Williams G, Larik A, Bok CW, Koh G, Clark RA. Modifiable Factors Associated With Poststroke Physical Activity at Discharge From Rehabilitation: Prospective Cohort Study. Phys Ther. 2020 May 18;100(5):818-828. doi: 10.1093/ptj/pzaa022. PMID 31995190
- [Background] Fini NA, Holland AE, Keating J, Simek J, Bernhardt J. How Physically Active Are People Following Stroke? Systematic Review and Quantitative Synthesis. Phys Ther. 2017 Jul 1;97(7):707-717. doi: 10.1093/ptj/pzx038. PMID 28444348
- [Background] Thilarajah S, Mentiplay BF, Bower KJ, Tan D, Pua YH, Williams G, Koh G, Clark RA. Factors Associated With Post-Stroke Physical Activity: A Systematic Review and Meta-Analysis. Arch Phys Med Rehabil. 2018 Sep;99(9):1876-1889. doi: 10.1016/j.apmr.2017.09.117. Epub 2017 Oct 19. PMID 29056502
- [Background] Moncion K, Biasin L, Jagroop D, Bayley M, Danells C, Mansfield A, Salbach NM, Inness E, Tang A. Barriers and Facilitators to Aerobic Exercise Implementation in Stroke Rehabilitation: A Scoping Review. J Neurol Phys Ther. 2020 Jul;44(3):179-187. doi: 10.1097/NPT.0000000000000318. PMID 32516297
- [Background] Committee for Proprietary Medicinal Products. Points to consider on switching between superiority and non-inferiority. Br J Clin Pharmacol. 2001 Sep;52(3):223-8. doi: 10.1046/j.0306-5251.2001.01397-3.x. No abstract available. PMID 11560553
- [Background] Yarnell CJ, Abrams D, Baldwin MR, Brodie D, Fan E, Ferguson ND, Hua M, Madahar P, McAuley DF, Munshi L, Perkins GD, Rubenfeld G, Slutsky AS, Wunsch H, Fowler RA, Tomlinson G, Beitler JR, Goligher EC. Clinical trials in critical care: can a Bayesian approach enhance clinical and scientific decision making? Lancet Respir Med. 2021 Feb;9(2):207-216. doi: 10.1016/S2213-2600(20)30471-9. Epub 2020 Nov 20. PMID 33227237
- [Background] Chang BH, Pocock S. Analyzing data with clumping at zero. An example demonstration. J Clin Epidemiol. 2000 Oct;53(10):1036-43. doi: 10.1016/s0895-4356(00)00223-7. PMID 11027937
- [Background] Thorn JC, Coast J, Cohen D, Hollingworth W, Knapp M, Noble SM, Ridyard C, Wordsworth S, Hughes D. Resource-use measurement based on patient recall: issues and challenges for economic evaluation. Appl Health Econ Health Policy. 2013 Jun;11(3):155-61. doi: 10.1007/s40258-013-0022-4. PMID 23529715
- [Background] Hodgson TA. Costs of illness in cost-effectiveness analysis. A review of the methodology. Pharmacoeconomics. 1994 Dec;6(6):536-52. doi: 10.2165/00019053-199406060-00007. PMID 10155283
- [Background] Stinnett AA, Mullahy J. Net health benefits: a new framework for the analysis of uncertainty in cost-effectiveness analysis. Med Decis Making. 1998 Apr-Jun;18(2 Suppl):S68-80. doi: 10.1177/0272989X98018002S09. PMID 9566468